CLINICAL TRIAL: NCT07021924
Title: The Effect of Fu's Subcutaneous Needling and Acupuncture on Local and Distal Skin Temperature in Healthy Subjects
Brief Title: The Effect of Fu's Subcutaneous Needling on Skin Temperature in Healthy Subjects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH113-REC1-151
Record Dates: First submitted 2025-04-20; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Skin Temperature Change
Keywords: Fu's subcutaneous needling; acupuncture; skin temperature; skin blood flow; hemodynamics
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fu's subcutaneous needling (Experimental): Fu's subcutaneous needling at acupoint LI-18
  Interventions: Other: Fu's subcutaneous needling
- Acupucture (Experimental): Acupuncture at acupoint LI-18
  Interventions: Other: Acupuncture
- Control (No Intervention): As the control group, Participants do not receive any intervention

INTERVENTIONS:
Other: Fu's subcutaneous needling — A single-use Fu's Subcutaneous Needling (FSN) device was employed. Participants were instructed to lie supine with the tested upper limb extended in a neutral position. After a 15-minute resting period, the FSN needle was fully inserted into the subcutaneous tissue layer at the acupoint Xialian (LI18) along the Large Intestine Meridian, with the needle tip oriented toward the radial styloid process.
  The needle core was retracted into the soft tube, and the needle was then manipulated by swinging the handle left and right in a fan-shaped manner, with a sweep angle of approximately 60 degrees (30 degrees in each direction) relative to the insertion axis. The swaying movements was performed 50 times back and forth (100 cycles/min) over a duration of 2 minutes.
  The needle was retained in place for 15 minutes before being removed. After needle removal, participants remained resting for 3 minutes before getting up, marking the end of the experimental procedure.
  Arms: Fu's subcutaneous needling
Other: Acupuncture — Participants were instructed to lie supine with the tested upper limb extended in a neutral position. According to WHO standard acupoint locations, the acupuncture needle was inserted at Xialian (LI18), located 4 cun below Quchi (LI11) on the line connecting Hegu (LI4) and Quchi (LI11). A 30-gauge, 1.5-inch acupuncture needle was used, and insertion continued until the Deqi sensation was achieved.
  The needle was retained for 15 minutes before being removed. After a 3-minute post-removal rest period, participants were allowed to rise, completing the procedure.
  Arms: Acupucture

SUMMARY:
The goal of this clinical trial is to investigate whether there are differences in skin temperature at local or distal sites following Fu's Subcutaneous Needling (FSN) treatment or acupuncture treatment, and compare the extent to which FSN or acupuncture induces an increase in skin temperature in healthy population. The main questions it aims to answer are:

1. Fu's Subcutaneous Needling (FSN) treatment increases local blood perfusion, thereby elevating skin temperature.
2. The ability of FSN treatment to increase skin temperature is not inferior to that of acupuncture and may, in fact, be superior.

Researchers will compare the skin temperature changes among three groups which are FSN, acupuncture and control group to see if there are statistically significantly changes .

Participants will enroll into three groups which are FSN, acupuncture and no any intervention respectively.

DETAILED DESCRIPTION:
Human physiological thermoregulation involves adjustments in heat dissipation and heat production in response to various internal and external thermal stimuli. The central control of thermoregulation is located in the preoptic/anterior hypothalamus (PO/AH) of the brain. Information about internal core and surface skin temperatures is transmitted to the PO/AH, which then coordinates appropriate responses. Skin blood flow is regulated by sympathetic nerve fibers, which release norepinephrine. When the core or surface temperature decreases, the intensity of sympathetic nerve activity increases, causing vasoconstriction at the arteriovenous anastomoses, resulting in reduced blood flow and decreased heat loss. Conversely, when the core or surface temperature increases, reduced sympathetic activity leads to vasodilation.

Numerous studies have utilized measurements of skin temperature and skin blood flow in traditional Chinese medicine research. Fu's subcutaneous needling therapy is widely used for treating conditions related to myofascial trigger points, as it is theorized to relieve the energy crisis that causes these trigger points by increasing blood perfusion in the affected muscles. However, fundamental research has not yet been completed to verify this theory. Therefore, this project aims to use skin temperature detection to determine whether Fu's subcutaneous needling can increase local skin blood perfusion and, compared to acupuncture, which method is more effective in raising skin temperature.

This study plans to recruit 60 healthy participants, who will be randomly assigned to the FSN group, acupuncture group, and control group. The participants will lie quietly in a temperature- and humidity-controlled room with nine detection points adhered to the right forearm. The entire experiment, including a 15-minute static phase, a 15-minute intervention phase, and a 3-minute post-intervention phase, will last 33 minutes. The researchers will record skin temperature every three minutes during the intervention and post-intervention phases, for a total of six recordings. Additionally, the investigator will measure changes in the hemodynamic parameters of the right forearm's radial artery using ultrasound before the static phase and after the post-intervention phase. Statistical analysis will be conducted on the changes in skin temperature at each detection point and hemodynamic parameters at radial artery.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participants aged 18 years or older, of any sex, who are able to fully comply with the experimental procedures.
* Recent medical examination confirming the absence of cardiovascular, respiratory, gastrointestinal, urinary, hematological, endocrine, and neurological disorders.
* Normal communication ability, with the capacity to understand and follow instructions related to Fu's Subcutaneous Needling (FSN) and acupuncture treatments.
* Provision of written informed consent.

Exclusion Criteria:

* Diagnosis of psychiatric disorders, severe depression, alcohol dependence, or a history of substance abuse.
* Pregnancy or breastfeeding.
* Presence of local skin infection, ulceration, or injury at the treatment site.
* Participation in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Skin Temperature | From enrollment to the end of treatment at 1 day
  Skin temperature was measured using the EXVXE® EX 3016 multi-channel temperature testing system (Yili [Shenzhen] Technology Co., Ltd.), which collects data from 16 thermistors affixed to the skin surface. Thermistors were attached to specific acupoints on the participants' right forearm along the Large Intestine Meridian of Hand-Yangming: Hegu (LI4), Yangxi (LI5), Pianli (LI6), Wenliu (LI7), Shousanli (LI10), and Quchi (LI11). Additional thermistors were placed on acupoints along the Small Intestine Meridian of Hand-Taiyang: Yanggu (SI5), Zhizheng (SI7), and Xiaohai (SI8).

SECONDARY OUTCOMES:
Hemodynamic Parameters: Peak Systolic Velocity (PSV, cm/s) | From enrollment to the end of treatment at 1 day
  Hemodynamic parameters were assessed using the Power Doppler (PD) mode of a GE LOGIQ e ultrasound system. Measurements were taken at the radial artery of the right arm, approximately one-quarter of the way up the forearm on the radial side.
  PSV:The maximum velocity of blood flow within a vessel during the systolic phase of the cardiac cycle, indicating the highest velocity achieved immediately following ventricular contraction.
Hemodynamic Parameters:End-Diastolic Velocity (EDV, cm/s) | From enrollment to the end of treatment at 1 day
  Hemodynamic parameters were assessed using the Power Doppler (PD) mode of a GE LOGIQ e ultrasound system. Measurements were taken at the radial artery of the right arm, approximately one-quarter of the way up the forearm on the radial side.
  EDV:The minimum velocity of blood flow measured at the end of cardiac diastole, reflecting the baseline velocity immediately before the subsequent ventricular contraction.
Hemodynamic Parameters: Mean Velocity (cm/s) | From enrollment to the end of treatment at 1 day
  Hemodynamic parameters were assessed using the Power Doppler (PD) mode of a GE LOGIQ e ultrasound system. Measurements were taken at the radial artery of the right arm, approximately one-quarter of the way up the forearm on the radial side.
  Mean Velocity:The average velocity of blood flow calculated over a specific cardiac cycle, representing the overall flow velocity across both systolic and diastolic phases.
Hemodynamic Parameters:Time-Averaged Mean Velocity (TAMV, cm/s) | From enrollment to the end of treatment at 1 day
  Hemodynamic parameters were assessed using the Power Doppler (PD) mode of a GE LOGIQ e ultrasound system. Measurements were taken at the radial artery of the right arm, approximately one-quarter of the way up the forearm on the radial side.
  TAMV:The mean velocity of blood flow averaged over multiple cardiac cycles, providing a representative steady-state measure of flow velocity.
Hemodynamic Parameters:Systolic/Diastolic Velocity Ratio (S/D) | From enrollment to the end of treatment at 1 day
  Hemodynamic parameters were assessed using the Power Doppler (PD) mode of a GE LOGIQ e ultrasound system. Measurements were taken at the radial artery of the right arm, approximately one-quarter of the way up the forearm on the radial side.
  S/D:A dimensionless ratio calculated by dividing the peak systolic velocity by the end-diastolic velocity, commonly used to evaluate arterial resistance and vascular compliance.
Hemodynamic Parameters:Arterial Diameter (d, cm) | From enrollment to the end of treatment at 1 day
  Hemodynamic parameters were assessed using the Power Doppler (PD) mode of a GE LOGIQ e ultrasound system. Measurements were taken at the radial artery of the right arm, approximately one-quarter of the way up the forearm on the radial side.
  d: The internal diameter of the artery at the measurement site, an essential parameter for calculating cross-sectional area, which directly influences flow calculations.
Hemodynamic Parameters:Resistance Index (RI) | From enrollment to the end of treatment at 1 day
  Hemodynamic parameters were assessed using the Power Doppler (PD) mode of a GE LOGIQ e ultrasound system. Measurements were taken at the radial artery of the right arm, approximately one-quarter of the way up the forearm on the radial side.
  RI: A dimensionless index calculated as (PSV - EDV)/PSV, quantifying arterial resistance and reflecting the vascular bed's impedance to blood flow.
Hemodynamic Parameters:Pulsatility Index (PI) | From enrollment to the end of treatment at 1 day
  Hemodynamic parameters were assessed using the Power Doppler (PD) mode of a GE LOGIQ e ultrasound system. Measurements were taken at the radial artery of the right arm, approximately one-quarter of the way up the forearm on the radial side.
  PI: A dimensionless index calculated as (PSV - EDV)/mean velocity, describing the pulsatile characteristics of arterial blood flow and providing insights into arterial elasticity and downstream vascular resistance.
Hemodynamic Parameters:Radial Artery Blood Flow (Q) | From enrollment to the end of treatment at 1 day
  Hemodynamic parameters were assessed using the Power Doppler (PD) mode of a GE LOGIQ e ultrasound system. Measurements were taken at the radial artery of the right arm, approximately one-quarter of the way up the forearm on the radial side.
  Q: Quantified as the volumetric blood flow rate (typically in cm³/s or ml/s), calculated by multiplying the vessel's cross-sectional area (derived from arterial diameter) by the time-averaged mean velocity (TAMV).

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided